## Effect of N-acetylcysteine on Exacerbations of Bronchiectasis (BENE): a randomized controlled trial

Official Title: Effect of N-acetylcysteine on Exacerbations of Bronchiectasis (BENE):

a randomized controlled trial

Trial registration: ClinicalTrials.gov (NCT02088216) (Registered date: March 5,

2014)

**Document Date:** November 2, 2018

## Statistical analyses

Patients who received at least one assessment visit after randomization were left in the original group for analysis of the results. Continuous data were expressed as the mean  $\pm$  standard deviation and were compared using the Student's t test. Categorical variables were expressed as a number (%) and were compared using the  $\chi^2$  test. Number of exacerbations was described by the median (interquartile range, IQR). The Mann-Whitney U test was performed to compare the difference in the number of exacerbations between the two groups. The primary study end point was the incidence of exacerbations, which is a count and follows Poisson distribution. Negative binomial regression not including other covariates was employed to compute the risk ratio and 95% confidence intervals (CIs) for N-acetylcysteine vs. the control. The time to the first exacerbation was described by Kaplan–Meier curves, and the log-rank test was used to explore the differences in time to the first exacerbation between the two groups. All analyses were conducted with the Statistical Package for the Social Sciences (SPSS) software (version 20.0). A p value < 0.05 was considered statistically significant.